CLINICAL TRIAL: NCT03804944
Title: Converting HR+ Breast Cancer Into an Individualized Vaccine
Acronym: CBCV
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Merck Sharp & Dohme LLC (Industry); Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1808019498
Record Dates: First submitted 2019-01-09; First posted 2019-01-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Patients will be on the study for a total of 5 months, this includes 4 months on active study intervention, with breast surgery at week 16 and one month follow up period, after surgery. Patients will be randomly assigned to one of the following arms. 1. Anti-PD1 antibody pembrolizumab (Keytruda, Merck) will be infused day 12, at the standard dose of 200 mg IV over 30 minutes, repeated every 3 weeks until disease progression or unacceptable toxicity. 2. FLT3L (CDX-301, the recombinant human protein by Celldex) will be self-administered subcutaneously, in 5 consecutive daily injections, week 1, day 1-5.
  3. For all arms radiation therapy to the breast tumor will begin on week 2 (Day 8,10,12), at dose of 8 Gy x 3 fractions, every other day. 4. Letrozole (Femara ®, Novartis) 2.5 mg tabs, once a day, daily for 4 months, until surgery, and thereafter is decided by the treating physician
Masking Description: Patients will be randomly assigned to one of the following arms. 1. Anti-PD1 antibody pembrolizumab (Keytruda, Merck) will be infused day 12, at the standard dose of 200 mg IV over 30 minutes, repeated every 3 weeks until disease progression or unacceptable toxicity. 2. FLT3L (CDX-301, the recombinant human protein by Celldex) will be self-administered subcutaneously, in 5 consecutive daily injections, week 1, day 1-5.
  3. For all arms radiation therapy to the breast tumor will begin on week 2 (Day 8,10,12), at dose of 8 Gy x 3 fractions, every other day. 4. Letrozole (Femara ®, Novartis) 2.5 mg tabs, once a day, daily for 4 months, until surgery, and thereafter is decided by the treating physician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- ARM 1 (Active Comparator): Focal hypo-fractionated radiation therapy 8 Gy x 3 fractions, starting day 8, every other day (M/W/F or W/F/M or F/M/W).
  Interventions: Radiation: Focal Radiation therapy
- ARM 2 (Active Comparator): Focal hypo-fractionated radiation therapy - 8 Gy x 3 fractions starting day 8, every other day (M/W/F or W/F/M or F/M/W). + Pembrolizumab, on day 12 (last day of radiotherapy), infused over 200mg IV over 30 minutes and then repeated every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Radiation: Focal Radiation therapy; Drug: Pembrolizumab (200mg IV for 30 minutes
- ARM 3 (Active Comparator): Ftl-3 ligand, self-administered by subcutaneous injections at week 1, daily, for 5 consecutive days + Focal hypo-fractionated radiation therapy - 8 Gy x 3 fractions starting day 8, (every other day (M/W/F or W/F/M or F/M/W).
  Interventions: Radiation: Focal Radiation therapy; Biological: CDX-301
- ARM 4 (Active Comparator): Ftl-3 ligand, self administered subcutaneous injections at day 1 for 5 consecutive days+ Focal hypo-fractionated Radiation therapy starting day 8, - 8 Gy x 3 fractions, every other day (M/W/F or W/F/M or F/M/W). + Pembrolizumab, on day 12 (last day of radiotherapy), 200mg IV infused over 30 minutes then repeated every 3 weeks until disease progression or unacceptable toxicity.
  Interventions: Radiation: Focal Radiation therapy; Drug: Pembrolizumab (200mg IV for 30 minutes; Biological: CDX-301

INTERVENTIONS:
Radiation: Focal Radiation therapy — Focal hypo-fractionated radiation therapy 8 Gy x 3 fractions, starting day 8, every other day (M/W/F or W/F/M or F/M/W).
Drug: Pembrolizumab (200mg IV for 30 minutes — Pembrolizumab, on day 12 (last day of radiotherapy), infused over 200mg IV over 30 minutes and then repeated every 3 weeks until disease progression or unacceptable toxicity.
  Arms: ARM 2; ARM 4
Biological: CDX-301 — Ftl-3 ligand, self-administered by subcutaneous injections at week 1, daily, for 5 consecutive days.
  Arms: ARM 3; ARM 4

SUMMARY:
Newly diagnosed post-menopausal women with clinical stage II-III, HR+HER2- breast cancer are eligible to a randomized trial, concurrently open at five US academic institutions. Patients receiving 4 months of standard neoadjuvant hormonal therapy with letrozole are randomly assigned to one of 4 arms of a trial testing focal hypo-fractionated RT alone or with immunotherapy combinations.

DETAILED DESCRIPTION:
Patients will be on the study for a total of 5 months, this includes 4 months on active study intervention, with breast surgery at week 16 and one month follow up period, after surgery. Patients will be randomly assigned to one of these 4 arms - 1. Anti-PD1 antibody pembrolizumab (Keytruda, Merck) will be infused day 12, at the standard dose of 200 mg IV over 30 minutes, repeated every 3 weeks until disease progression or unacceptable toxicity. 2. FLT3L (CDX-301, the recombinant human protein by Celldex) will be self-administered subcutaneously, in 5 consecutive daily injections, week 1, day 1-5. 3. For all arms radiation therapy to the breast tumor will begin on week 2 (Day 8,10,12), at dose of 8 Gy x 3 fractions, every other day. 4. Letrozole (Femara ®, Novartis) 2.5 mg tabs, once a day, daily for 4 months, until surgery, and thereafter is decided by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal female ≥ 18 years of age (Post-menopausal status defined as either 1) at least 2 years without menstrual period or 2) or patients older than 50 with serological evidence of post-menopausal status or 3) hysterectomized patients of any age with FSH confirmation of post-menopausal status.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Biopsy proven diagnosis of ER+ PR+ or PR- HER2- breast cancer.
* Clinical stage I(>1.5cm, if N0) - III breast cancer, as per AJCC staging 8th edition.
* Patient needs to be able to understand and demonstrate willingness to sign a written informed consent document.

Adequate bone marrow reserve and liver function:

WBC ≥ 2000/uL Absolute neutrophil count (ANC) ≥1500/μL Platelets ≥100 000/μL Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La Creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN AST (SGOT) and ALT (SGPT) ≤2.5 × ULN (≤5 × ULN for participants with liver metastases) International normalized ratio (INR) OR prothrombin time (PT) Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Active connective tissue disorders, such as lupus or scleroderma requiring flare therapy
* Current use of systemic chemotherapy, endoctine therap or HER2-neu targeted therapy
* Post surgical excision of breast cancer.
* Previous radiotherapy of the same breast.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
* Inability to obtain histologic proof of breast cancer
* Has received a live vaccine within 30 days prior to the first dose of study drug.

Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.

* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy (second primary) that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.Has a known history of Human Immunodeficiency Virus (HIV). Note: No HIV testing is required unless mandated by local health authority.
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis). Note: optional based on country.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Newly diagnosed postmenopausal patients with clinical stage I-III ER+HER- invasive breast cancer will be eligible to participate in this trial. Patients with invasive ductal or lobular or mixed ductal/lobular breast cancers are eligible. (Clinical Stage 1 tumor size - >1.5cm, if N0)
Enrollment: 100 (Estimated)
Dates: Start 2020-03-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerability will be demonstrated if no grade 3 or higher toxicities are observed in the first 8 patients, of each arm. | 3 years
  Tolerability of adding immunotherapy to a combination of tumor radiotherapy and endocrine therapy in the neoadjuvant setting of newly diagnosed HR+ breast cancer patients will be assessed if no grade 3 or higher toxicities are observed in the first 8 patients of each arm. CTCAE version 5.0 will be used.
Clinical response rate to tumor radiation +/-immunotherapy during standard endocrine therapy for HR+ breast cancer will be measured. | 3 years
  Clinical response rate to tumor radiation +/-immunotherapy during standard endocrine therapy for HR+ breast cancer will be measured.
Pathological response rate to tumor radiation +/-immunotherapy during standard endocrine therapy for HR+ breast cancer will be measured. | 3 years
  Pathological response rate to tumor radiation +/-immunotherapy during standard endocrine therapy for HR+ breast cancer will be measured.

SECONDARY OUTCOMES:
Local immune response will be measured by assessing tumor specimens for T-cell infiltration at baseline and and during treatment. | 4 years
  Local immune response will be measured by assessing tumor specimens for T-cell infiltration at baseline and and during treatment.
Systemic immune response will be measured by collecting serial blood samples for serum and peripheral blood mononuclear cells (PBMCs) at multiple time points. | 4 years
  Systemic immune response will be measured by collecting serial blood samples for serum and peripheral blood mononuclear cells (PBMCs) at multiple time points.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Formenti, M.D., Principal Investigator — Weill Cornell Medicine - New York Presbyterian Hospital
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Icahn School of Medicine at Mt Sinai, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York
  - Weill Cornell Medicine New York Presbyterian Hospital, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No